CLINICAL TRIAL: NCT06030674
Title: Measuring Environmental Tobacco and Cannabis: Pollutants and Exposures
Acronym: CAN03
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T32IR4867
Record Dates: First submitted 2023-08-25; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Nonsmokers; Secondhand cannabis smoke; Environmental cannabis; Exposure
MeSH Terms: interventions — Smoke

STUDY DESIGN:
Intervention Model Description: This is an unblinded pilot study of an environmental exposure in one group.
Masking Description: The exposure cannot be masked or blinded. Data analysts and chemists will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure to secondhand cannabis smoke in public places (Experimental): The research staff and participants will travel together to a public location by either ride share vehicles, taxis or public transit. The study will arrange and pay for the transit. Staff and participants will be exposed to ambient air in public places where cannabis products are being consumed by smoking, vaporizing or dabbing. Participants will remain in the company of the laboratory staff throughout the exposure. The exposures will last 0.5-4 hours, depending on the nature and duration of the event. Staff and participants will travel together back to the laboratory for the post-exposure study measures.
  Interventions: Other: Secondhand cannabis emissions/smoke exposure

INTERVENTIONS:
Other: Secondhand cannabis emissions/smoke exposure — This is an environmental exposure performed in public places where people are consuming cannabis.

SUMMARY:
This is an unblinded pilot study of an environmental exposure to secondhand cannabis smoke in one group of healthy nonsmokers.

DETAILED DESCRIPTION:
The goal is to gather accurate information on uptake of smoke toxicants from cannabis exposures in the real world. The investigators will be taking healthy nonsmokers to public places where people are consuming cannabis and measuring their uptake of cannabinoids.

ELIGIBILITY:
Inclusion Criteria:

-

Adult nonsmokers, aged 21-50, who:

* Are healthy on the basis of medical history
* Have systolic blood pressure <150
* Have diastolic blood pressure <100
* Have BMI between 18.1 and 34.9
* Able to perform moderate exercise,
* Are not exposed to tobacco or cannabis SHS in their daily lives. (Nonsmoking status and low SHS exposure are determined by self-report on the screening questionnaire, salivary cotinine < 10 ng/ml and THC < 50 ng/m and exhaled CO2 below 4 ppm)

Exclusion Criteria:

* Current use of cannabis products, including CBD and edible THC products
* Regular exposure to secondhand tobacco or cannabis smoke
* Positive SARS-CoV-2 antibody test
* Age 18 < or > 50
* Physician diagnosis of asthma, heart disease, hypertension, thyroid disease, diabetes, renal or liver impairment or glaucoma.
* Unstable psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder) or current use of more than two psychiatric medications
* Systolic blood pressure > 150
* Diastolic blood pressure > 100
* Pregnancy or breastfeeding (by urine hCG and/or history)
* Alcohol or illicit drug dependence within the past 5 years
* BMI > 35 and < 18
* Current illicit drug use (by history or urine test)
* More than 1 pack year smoking history
* Ever a daily marijuana smoker
* Smoked anything within the last 2 months
* Occupational exposure to smoke, dusts OR fumes
* Concurrent participation in another clinical trial
* Unable to communicate in English
* No social security number

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the concentration of urinary cannabinoid metabolites in health nonsmokers exposed to cannabis smoke and emissions | Baseline (before exposure) and the morning after exposure, up to 22 hours.
  The concentration of 11-Nor-9-carboxy-THC will be measured in urine with LC/MS-MS. The LOQ for this assay is 15 pg/ml. Anticipated changes in concentration are from BLOQ to 0.5-20 ng/ml. The duration of the exposures will depend on the event or venue at which exposures occur, ranging from 30 minutes to 4 hours. The investigators will compare the concentration of 11-Nor-9-carboxy-THC in participants' urine before exposure to concentrations in the first void of the morning after the day of exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Suzaynn F Schick, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No